CLINICAL TRIAL: NCT00140049
Title: A 12-Week Randomized, Evaluator-Masked, Parallel-Group, Multinational, Multi-Center Study Comparing The Efficacy And Safety Of The Fixed Combination Of Latanoprost And Timolol (Xalacom) With The Fixed Combination Of Dorzolamide And Timolol (Cosopt) In Patients With Open-Angle Glaucoma Or Ocular Hypertension.
Brief Title: A 12week, Randomized, Evaluator-Masked, Parallel Group Comparing Evening Dosing Of Xalacom Vs Cosopt In Subj W/ Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A6641038
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2007-11

CONDITIONS: Glaucoma, Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Xalacom; dorzolamide-timolol combination

INTERVENTIONS:
Drug: Xalacom
Drug: Cosopt

SUMMARY:
To demonstrate the statistical non inferiority of the combination of latanoprost and timolol given in the evening time once a day vs the combination of dorzamalide and timolol twice a day based on intraocular pressure measurements at 8 AM, 12 noon & 4 PM during a 12 week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral diagnosis of primary open angle glaucoma or ocular hypertension on beta-blocker monotherapy or dual therapy in which at least one medication is a beta-blocker for at least 4 weeks prior to screening

Exclusion Criteria:

* Closed/ barely open anterior chamber angle or history of acute angle closure glaucoma.
* History of ALT (Argon Laser Trabeculoplasty) or SLT(selective Laser) within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238
Dates: Start 2005-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The mean IOP measurements obtained in the study eye at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- France (5):
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Saint-Herblain
- Germany (5):
  - Pfizer Investigational Site, Darmstadt
  - Pfizer Investigational Site, Landau / Pfalz
  - Pfizer Investigational Site, Regenstauf
  - Pfizer Investigational Site, Schorndorf
  - Pfizer Investigational Site, Starnberg
- Greece (4):
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Thessaloniki, Macedonia
  - Pfizer Investigational Site, Alexandroupoli
  - Pfizer Investigational Site, Larissa
- Italy (6):
  - Pfizer Investigational Site, Chieti
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Monza (MI)
  - Pfizer Investigational Site, Pisa
- Sweden (4):
  - Pfizer Investigational Site, Ã¶rebro
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Sundsvall